CLINICAL TRIAL: NCT04652648
Title: Rapid Development and Implementation of a Remote ECG-monitored Prospective Randomized Clinical Trial During a Pandemic: Hydroxychloroquine Prophylaxis in COVID-19 Household Contacts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bryn Mawr Hospital (Other)
Collaborators: Sharpe-Strumia Research Foundation (Other); Bryn Mawr Hospital Foundation (Unknown); Cotswold Foundation (Unknown)
Responsible Party: Principal Investigator, Luciano kapelusznik, Attending Physician, Bryn Mawr Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BM02332
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Covid19; Hydroxychloroquine; Coronavirus Infection; Transmission; Prophylaxis
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): Randomization was 2:1 to HCQ 200 mg BID for 10 days
  Interventions: Drug: Hydroxychloroquine
- Control (No Intervention): No Intervention

INTERVENTIONS:
Drug: Hydroxychloroquine — Randomization was 2:1 to HCQ 200 mg BID or 41 observation for 10 days
  Arms: Hydroxychloroquine

SUMMARY:
* organizing an entirely no in-person contact clinical trial is feasible during a 22 COVID-19 pandemic 23
* Remote smartphone 6-lead ECG monitoring is possible even in a group unfamiliar 24 with the technology 25
* Hydroxychloroquine used prophylactically at 200 mg BID had no observable 26 cardiotoxicity 27
* Additional study using this technique is warranted to look at reliability and cost-28 effectiveness

DETAILED DESCRIPTION:
Household members were contacted by telephone and provided consent forms via E-mail electronic signatures. Randomization was 2:1 to HCQ 200 mg BID or observation for 10 days with total follow-up of 14 days. COVID status was determined by home saliva PCR assay on days 1 and 14. Study drug was shipped to participants. Data of daily symptoms and 6-lead ECGs using a smartphone KardiaMobile® 6L application were collected.

ELIGIBILITY:
Inclusion Criteria:

* exposure to a COVID-19-infected individual in the same household within five days of diagnosis;
* age >18 years;
* ability to give informed consent to participate in a clinical study;
* ability to swallow oral medications;
* access to a smartphone

Exclusion Criteria:

* allergy or intolerance to hydroxychloroquine (PlaquenilR);
* weight less than 85 pounds;
* eye disease affecting the retina;
* severe kidney or liver disease;
* G6PD-deficiency;
* porphyria;
* long QTc EKG abnormality or family history of this;
* other major EKG abnormalities;
* taking medications that can affect the QT interval including flecainide, amiodarone, digoxin, procainamide, propafenone, sotalol, quinidine, dofetilide, levofloxacin, ciprofloxacin, azithromycin, erythromycin, amitriptyline, doxepin, desipramine, imipramine, fluoxetine, sertraline, venlafaxine, quetiapine, haloperidol, droperidol, thioridazine, ziprasidone, furosemide, sumatriptan or zolmitriptan, cisapride, arsenic, dolasetron, or methadone;
* current pregnancy;
* current hospitalization;
* symptomatic with fever or cough;
* lack of access to a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
COVID-19 symptom development with positive PCR test | within 14 days
  The primary endpoint was development of COVID-19 symptoms with a positive coronavirus PCR test by Day 14.

SECONDARY OUTCOMES:
Positive coronavirus PCR test without symptoms | By Day 14 (end of study)
  Development of a positive coronavirus PCR test without symptoms by Day 14
Hospital admission for COVID-19 | within 14 days of study entry
  hospital admission for COVID-19 symptoms by Day 14
Death by Day 14 | within 14 days of study entry
  Death due to COVID-19 within 14 days of study entry
HCQ discontinuation or study withdrawal | within 14 days of study entry
  All-cause discontinuation of study medication or study withdrawal by Day 14
Symptom severity at specified time points | at Day 7 and at Day 14 from study entry
  overall symptom severity at Day 7 and Day 14
COVID -19 rate at study entry | Day 1 of study
  household attack rate at study entry
EKG changes during study | Day 1 thru Day 14 of study
  documentation of EKG changes such as QTc prolongation on HCQ compared with no drug therapy

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Background] Lauer SA, Grantz KH, Bi Q, Jones FK, Zheng Q, Meredith HR, Azman AS, Reich NG, Lessler J. The Incubation Period of Coronavirus Disease 2019 (COVID-19) From Publicly Reported Confirmed Cases: Estimation and Application. Ann Intern Med. 2020 May 5;172(9):577-582. doi: 10.7326/M20-0504. Epub 2020 Mar 10. PMID 32150748
- [Background] Day M. Covid-19: identifying and isolating asymptomatic people helped eliminate virus in Italian village. BMJ. 2020 Mar 23;368:m1165. doi: 10.1136/bmj.m1165. No abstract available. PMID 32205334
- [Background] Rolain JM, Colson P, Raoult D. Recycling of chloroquine and its hydroxyl analogue to face bacterial, fungal and viral infections in the 21st century. Int J Antimicrob Agents. 2007 Oct;30(4):297-308. doi: 10.1016/j.ijantimicag.2007.05.015. Epub 2007 Jul 16. PMID 17629679
- [Background] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Background] Colson P, Rolain JM, Lagier JC, Brouqui P, Raoult D. Chloroquine and hydroxychloroquine as available weapons to fight COVID-19. Int J Antimicrob Agents. 2020 Apr;55(4):105932. doi: 10.1016/j.ijantimicag.2020.105932. Epub 2020 Mar 4. No abstract available. PMID 32145363
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Mitja O, Clotet B. Use of antiviral drugs to reduce COVID-19 transmission. Lancet Glob Health. 2020 May;8(5):e639-e640. doi: 10.1016/S2214-109X(20)30114-5. Epub 2020 Mar 19. No abstract available. PMID 32199468
- [Background] Vincent MJ, Bergeron E, Benjannet S, Erickson BR, Rollin PE, Ksiazek TG, Seidah NG, Nichol ST. Chloroquine is a potent inhibitor of SARS coronavirus infection and spread. Virol J. 2005 Aug 22;2:69. doi: 10.1186/1743-422X-2-69. PMID 16115318
- [Background] Principi N, Esposito S. Chloroquine or hydroxychloroquine for prophylaxis of COVID-19. Lancet Infect Dis. 2020 Oct;20(10):1118. doi: 10.1016/S1473-3099(20)30296-6. Epub 2020 Apr 17. No abstract available. PMID 32311322
- [Background] Marquis-Gravel G, Roe MT, Turakhia MP, Boden W, Temple R, Sharma A, Hirshberg B, Slater P, Craft N, Stockbridge N, McDowell B, Waldstreicher J, Bourla A, Bansilal S, Wong JL, Meunier C, Kassahun H, Coran P, Bataille L, Patrick-Lake B, Hirsch B, Reites J, Mehta R, Muse ED, Chandross KJ, Silverstein JC, Silcox C, Overhage JM, Califf RM, Peterson ED. Technology-Enabled Clinical Trials: Transforming Medical Evidence Generation. Circulation. 2019 Oct 22;140(17):1426-1436. doi: 10.1161/CIRCULATIONAHA.119.040798. Epub 2019 Oct 21. PMID 31634011
- [Background] Turakhia MP, Desai M, Hedlin H, Rajmane A, Talati N, Ferris T, Desai S, Nag D, Patel M, Kowey P, Rumsfeld JS, Russo AM, Hills MT, Granger CB, Mahaffey KW, Perez MV. Rationale and design of a large-scale, app-based study to identify cardiac arrhythmias using a smartwatch: The Apple Heart Study. Am Heart J. 2019 Jan;207:66-75. doi: 10.1016/j.ahj.2018.09.002. Epub 2018 Sep 8. PMID 30392584
- [Background] Spaccarotella CAM, Polimeni A, Migliarino S, Principe E, Curcio A, Mongiardo A, Sorrentino S, De Rosa S, Indolfi C. Multichannel Electrocardiograms Obtained by a Smartwatch for the Diagnosis of ST-Segment Changes. JAMA Cardiol. 2020 Oct 1;5(10):1176-1180. doi: 10.1001/jamacardio.2020.3994. PMID 32865545
- [Derived] Liu HH, Ezekowitz MD, Columbo M, Khan O, Martin J, Spahr J, Yaron D, Cushinotto L, Kapelusznik L. The future is now: our experience starting a remote clinical trial during the beginning of the COVID-19 pandemic. Trials. 2021 Sep 7;22(1):603. doi: 10.1186/s13063-021-05537-6. PMID 34493311
- [Derived] Liu HH, Ezekowitz MD, Columbo M, Khan O, Martin J, Spahr J, Yaron D, Cushinotto L, Kapelusznik L. Testing the feasibility of operationalizing a prospective, randomized trial with remote cardiac safety EKG monitoring during a pandemic. J Interv Card Electrophysiol. 2022 Mar;63(2):345-356. doi: 10.1007/s10840-021-00989-x. Epub 2021 May 26. PMID 34037911